CLINICAL TRIAL: NCT05947864
Title: Monitoring of Measles-specific Immune Status in Adult Allogeneic Hematopoietic Stem Cell Transplant Recipients: a Prospective Cohort Study
Brief Title: Monitoring of Measles-specific Immune Status in Adult Allogeneic Hematopoietic Stem Cell Transplant Recipients
Acronym: MaRROwVacc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0364; 2023-A00901-44 (Other: ID RCB)
Record Dates: First submitted 2023-06-28; First posted 2023-07-17 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Transplantation, Hematopoietic Stem Cell
MeSH Terms: interventions — Blood Specimen Collection; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allo-HSCT recipients (Experimental): Adult recipients of allogenic hematopoietic stem cell transplantation, eligible for live-attenuated vaccines, i.e. who are more than 24 months after their HSCT, without GVHD and more than 3 months after cessation of any immunosuppressant treatment
  Interventions: Biological: Biological samples (blood and oral fluid)
- Healthy volunteers (HV) (Placebo Comparator): Healthy adults with a history of measles (=convalescents) or vaccinated with two doses of MMR in the past (=vaccinated)
  Interventions: Biological: Biological samples (blood and oral fluid)

INTERVENTIONS:
Biological: Biological samples (blood and oral fluid) — For the study population (allo-HSCT recipients): 4 visits with biological sampling (blood and oral fluid) at each visit:
  * Visit V1 (inclusion visit = D1): immediately before the first dose of MMR (dose-1),
  * Visit V2 (D1 + 35 (+/-7) days): immediately before the second dose of MMR (dose-2)
  * Visit V3 (D1 + 70 (+/-14) days)
  * Visit V4 (D1 + 365 (+/-90) days) For healthy volunteers: a single visit (V1) with biological sampling (blood and oral fluid)

SUMMARY:
Measles, a highly contagious disease, is potentially serious in adult allogenic hematopoietic stem cell transplant (allo-HSCT) recipients. Because of the loss of immunity to vaccine preventable diseases after allo-HSCT, French Health Authorities (Haut Conseil de Santé Publique, HCSP) recommend (re)vaccination of all allo-HSCT recipients against measles-mumps-rubella (MMR) from 24 months post-transplant onwards, in the absence of graft-versus-host disease (GVHD) and at least 3 months after cessation of all immunosuppressive treatments, irrespective of measles serostatus. Nevertheless, some French experts argue that systematic assessment of measles antibody titre is justified after allo-HSCT, prior to revaccination, in order to avoid "unnecessary" revaccination of allo-HSCT recipients who are still seropositive. At the international level, recommendations also vary: the ECIL group and IDSA advocate revaccination of measles seronegative patients only, while some American Hematology experts recommend not to base the decision of revaccination on the serological status, given the inevitable loss of antibodies and specific long-term immune memory in the absence of revaccination.

Several obstacles to the application of the recommendations can therefore be identified: (i) the risk of vaccine-transmitted disease due to the live-attenuated nature of MMR, (ii) the lack of robust data on the immunogenicity and tolerability of the MMR vaccine in this particular population, and (iii) conflicting recommendations to guide the decision of revaccination.

This study aims at answering the question of whether some allo-HSCT recipients may retain a measles-specific cellular immune memory at distance from their allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

Study population:

* Aged ≥ 18 years and ≤ 75 years,
* Have received an allo-HSCT ≥ 24 months ago,
* In complete remission of initial hematologic disease and with successful engraftment (recipient chimerism <0.3% on whole blood),
* Without extensive chronic GVHD,
* Having given their written consent,
* Affiliated to a social security plan,
* Able to attend all scheduled visits and to comply with all study procedures.

Healthy volunteers:

* Aged ≥ 18 years and ≤ 75 years,
* Having a history of measles (=convalescent) or have been vaccinated in the past with two doses of MMR (=vaccinated),
* Having given their written consent,
* Affiliated to a social security plan.

Exclusion Criteria:

Study population:

* History of autoimmune disease or acquired immunodeficiency (other than the hematological disease),
* Patients undergoing pharmacological immunosuppression or biotherapy or extracorporeal photopheresis at the time of inclusion, or whose immunosuppressive treatment (corticosteroids and anti-rejection agents) has been stopped less than 3 months ago, or whose biotherapy (anti-cytokines, anti-JAK, anti-CD20 etc.) has been stopped less than 3 months ago (12 months for anti-CD20 including rituximab), or whose extracorporeal photopheresis has been stopped less than 3 months ago,
* Patients having received ≥ 1 infusion of IVIG in the 8 months prior to inclusion,
* Patients whose last HSCT was an autograft,
* Patients with known chronic active infection with human immunodeficiency virus (HIV) and/or hepatitis B or C virus(es),
* Patients deprived of liberty by judicial or administrative decision,
* Patients under legal protection or unable to consent to the study,
* Patients participating in another interventional research study with an exclusion period still in progress at pre-inclusion,
* Pregnant, parturient or breast-feeding women.

Healthy volunteers:

* History of autoimmune disease or acquired immunodeficiency,
* History of pharmacological immunosuppression or biotherapy discontinued less than 3 months ago (12 months for anti-CD20 including rituximab),
* History of IVIG infusion in the 8 months prior to inclusion,
* Persons deprived of liberty by judicial or administrative decision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Combined quantification of measles-specific markers of T-cell-mediated immunity (interferon-gamma [IFNγ]-secreting cells; copies of ifnγ mRNA transcripts; amount of IFNγ) and B-cell-mediated immunity (antibody-secreting cells [ASC]) | At Day 1, before routine vaccination with MMR in allo-HSCT recipients
  To explore the measles-specific T- and B-cell-mediated systemic immune memory pre-existing to MMR (re)vaccination in allo-HSCT recipients eligible for MMR revaccination according to current French recommendations (i.e., regardless of measles serostatus), T- and B-ELISpot techniques on PBMC, qPCR and cytokine measurement on whole blood, will be performed after ex vivo antigen stimulation

SECONDARY OUTCOMES:
Kinetics of anti-measles total IgG and IgA titers (serum) | At Day 1, Day 35, Day 70 and Day 365 in allo-HSCT recipients
  To characterize the total measles-specific systemic humoral immune response before and after MMR (re)vaccination, anti-measles antibodies will be measured in serum by ELISA
Kinetics of anti-measles neutralizing antibody titers (serum) | At Day 1, Day 70 and Day 365 in allo-HSCT recipients
  To characterize the neutralizing measles-specific systemic humoral immune response before and after MMR (re)vaccination, neutralizing serum antibodies titers will be determined through seroneutralization techniques
Combined quantification of measles-specific markers of T-cell-mediated immunity (IFNγ-secreting cells; copies of ifnγ mRNA transcripts; amount of IFNγ) and B-cell-mediated immunity (ASC) after two doses of MMR | At Day 365, after completion of MMR (re)vaccination schedule in allo-HSCT recipients
  To explore the measles-specific T- and B-cell-mediated systemic immune response after completing MMR (re)vaccination, T- and B-ELISpot techniques on PBMC, qPCR and cytokine measurement on whole blood, will be performed after ex vivo antigen stimulation
Kinetics of anti-measles IgA titers (oral fluid) | At Day 1 and Day 70 in allo-HSCT recipients
  To characterize the measles-specific mucosal humoral immune response before and after MMR (re)vaccination, anti-measles IgA will be measured in oral fluid by ELISA
Difference in immunity markers (total IgG and IgA, neutralizing antibody titers [serum]; IgA titers [oral fluid]; IFNγ-secreting cells; copies of ifnγ mRNA transcripts; amount of IFNγ; ASC) between HV and allo-HSCT recipients | At Day 1 and Day 70
  To compare the measles-specific systemic and mucosal immune response between convalescent/vaccinated HV and allo-HSCT recipients, markers of B-cell and T-cell-mediated immunity will be evaluated in convalescent/vaccinated HV at a single timepoint and compared to immunity markers evaluated in allo-HSCT recipients before and after MMR (re)vaccination
Analysis of measles-specific immunity markers (total IgG and IgA, neutralizing antibody titers [serum]; IgA titers [oral fluid]; IFNγ-secreting cells; copies of ifnγ mRNA transcripts; amount of IFNγ; ASC) according to patient characteristics | At Day 1, Day 35, Day 70 and Day 365 in allo-HSCT recipients
  To determine the impact of demographic, hematological, transplant-related characteristics, post-transplant complications and measles serostatus on measles-specific B-cell and T-cell immunity markers, before and after MMR (re)vaccination, bivariate and multivariate analysis will be carried out
Local and systemic adverse events after the first and the second MMR dose | At Day 35 and Day 70, in allo-HSCT recipients
  To describe the tolerance of the two MMR schedule in allo-HSCT recipients, solicited adverse events will be recorded up to day+14 and unsolicited adverse events will be recorded up to day+28 after each MMR dose through self-monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Anne CONRAD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse - service des maladies infectieuses et tropicales, Lyon, France